CLINICAL TRIAL: NCT05557682
Title: Clinical Performance and Psychological Impact of Colored Poly-acid Modified Composite Resin Versus Glass Ionomer Cement in Primary Molars: an RCT Study
Brief Title: Clinical Performance and Psychological Impact of Colored Restorations Cement in Primary Molars
Status: Completed | Type: Observational
Sponsor: British University In Egypt (Other)
Responsible Party: Principal Investigator, Nadia Metwalli, Professor of Pediatric Dentistry, British University In Egypt
Other Study IDs: FDBUEREC21-30
Record Dates: First submitted 2022-02-02; First posted 2022-09-28 (Actual); Last update posted 2022-09-28 (Actual); Status verified 2022-09

CONDITIONS: Pediatric Dentistry

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- clinical performance: restoration of caries primary molars using two different restorative materials
  Interventions: Other: composite restorative treatment
- psychological impact: evaluation of colour of restoration on the satisfaction of the children and impact on their hygiene

INTERVENTIONS:
Other: composite restorative treatment — Restorative treatment using dental materials
  Other Names: glass ionomer restorative treatment
  Groups: clinical performance

SUMMARY:
Aim of the study

The aim of the presented study is to evaluate:

I- The clinical performance of flowable polyacid-modified composite resin 'compomer' and resin-modified glass-ionomer cement in prepared Class II cavities in primary molars over a period of 6 months.

II- Psychological impact of the coloured material used on the child's behavior towards the dental procedure.

Materials and Methods Forty primary molars from healthy children between ages of four and seven years will be included in this study, parents will be asked to sign an informed consent on behalf of the children. Statistical power analysis was performed using G-power program. An alpha type error of 0.05, a beta power of 0.95 and a N2/N1 ratio of 1 was used. This study have the approval of the research ethics committee BUE. This study will be executed in the Faculty of Dentistry, BUE, Department of Pediatric Dentistry. Subjects will be selected from children who are seeking dental treatment at the Pediatric Dentistry and Dental Public Health clinic in the Faculty of Dentistry, BUE. Children with detectable caries for Class II cavity preparation will be classified randomly under the different treatment groups. Group A: Colored polyacid modified composite resin , Group B: Glass ionomer cement All groups will be restored according to material used. Restorations will be assessed for marginal adaptation, marginal discoloration, anatomic form, and secondary caries. The assessment of all restorations will be carried out at 24-hours, 3, 6 months post-operatively under normal clinical conditions with a dental operating light, a mouth mirror and a dental explorer. The impact of the color of the material used on the child's attitude will be assessed once through a questionnaire given to the child at the beginning of the first dental visit in which each child will be asked to choose from pictures that indicate their preference regarding the use of colored and non-colored restorative materials and how their choice will affect their attitude whether they will be happy, sad or neutral.

As per the scheduled follow up visits, these are the regular follow up intervals for any child undergoing dental treatment. Accordingly, it won't be of an extra burden on the patient/ parent.

Statistical analysis Data will be collected, tabulated and statistically analyzed using statistical package for Social Science (SPSS 15.0.1 for windows; SPSS Inc, Chicago, IL, 2001). Data will be presented and suitable analysis will be done according to the type of data obtained for each parameter.

DETAILED DESCRIPTION:
Aim of the study

The aim of the presented study is to evaluate:

I- The clinical performance of flowable polyacid-modified composite resin 'compomer' and resin-modified glass-ionomer cement in prepared Class II cavities in primary molars over a period of 6 months.

II- Psychological impact of the coloured material used on the child's behavior towards the dental procedure.

Materials and Methods Forty primary molars from children between ages of four and seven years will be included in this study, parents will be asked to sign an informed consent on behalf of the children. Statistical power analysis was performed using G-power program. An alpha type error of 0.05, a beta power of 0.95 and a N2/N1 ratio of 1 was used. This study will have the approval of the research ethics committee BUE and will be registered in clinical trial website.

This study will be executed in the Faculty of Dentistry, ,BUE,Department of Pediatric Dentistry. Subjects will be selected from children who are seeking dental treatment at the Pediatric Dentistry and Dental Public Health clinic in the Faculty of Dentistry, BUE. Children with detectable caries for Class II cavity preparation will be classified randomly under the different treatment groups.

Group A: Colored polyacid modified composite resin Group B: Glass ionomer cement

Children will be recruited according to the following inclusion and exclusion criteria:

Table 1: Inclusion and exclusion criteria Inclusion criteria Exclusion criteria Radiographic examination (bite-wing radiograph) showing evidence of proximal caries. Radiographic examination (bite-wing radiograph) showing evidence of occlusal caries only, or showing evidence of proximal caries extending to the pulp.

Proximal contact with adjacent healthy or restored tooth. Isolated tooth No signs or symptoms of pulp involvement Signs or symptom of pulp involvement.

No signs of periapical pathosis Signs of periapical pathosis No signs of periodontal involvement Signs of periodontal involvement 2 years at least till normal exfoliation Less than 2 years for exfoliation 2/3 of the root is still present Less than 2/3 of the root is present No restoration present Restoration present No cuspal involvement Cuspal involvement

All groups will be restored according to material used. Restorations will be assessed for marginal adaptation, marginal discoloration, anatomic form, and secondary caries. The assessment of all restorations will be carried out at 24-hours, 3, 6 months post-operatively under normal clinical conditions with a dental operating light, a mouth mirror and a dental explorer.

The impact of the color of the material used on the child's attitude will be assessed once through a questionnaire given to the child at the beginning of the first dental visit in which each child will be asked to choose from pictures that indicate their preference regarding the use of colored and non-colored restorative materials and how their choice will affect their attitude whether they will be happy, sad or neutral.

It is worth mentioning that the children selected for this study will be given meticulous oral hygiene measures instructions and will undergo full dental treatment during the course of the study thus, there are absolutely no risks on the human participants especially that only the decayed molars will be filled using the two different materials used in this study. However, chances of loss of the filling material, secondary caries, loss of the anatomical form, marginal discolouration and loss of the marginal adaptation might still be a subject of concern.

If these materials have been proved to be durable, more accepted by the children and less technique sensitive to the clinician then the patient/parent will be informed by the results and given the choice in case he/she wishes to change the restoration at any point and time.

As per the scheduled follow up visits, these are the regular follow up intervals for any child undergoing dental treatment. Accordingly, it won't be of an extra burden on the patient/ parent.

Statistical analysis Data will be collected, tabulated and statistically analyzed using statistical package for Social Science (SPSS 15.0.1 for windows; SPSS Inc, Chicago, IL, 2001). Data will be presented and suitable analysis will be done according to the type of data obtained for each parameter.

1. Descriptive Statistics: frequency and percentage of non-numerical data
2. Analytical Statistics: The Cochran Q procedure tests the null hypothesis that multiple related proportions are the same. The Cochran test is a multivariate extension of the McNemar test used for two related samples.

ELIGIBILITY:
Inclusion Criteria:

* Radiographic examination (bite-wing radiograph) showing evidence of proximal caries.
* Proximal contact with adjacent healthy or restored tooth.
* No signs or symptoms of pulp involvement
* No signs of periapical pathosis
* No signs of periodontal involvement
* 2 years at least till normal exfoliation
* 2/3 of the root is still present
* No restoration present
* No cuspal involvement

Exclusion Criteria:

* Radiographic examination (bite-wing radiograph) showing evidence of occlusal caries only, or showing evidence of proximal caries extending to the pulp.
* Isolated tooth
* Signs or symptom of pulp involvement.
* Signs of periapical pathosis
* Signs of periodontal involvement
* Less than 2 years for exfoliation
* Less than 2/3 of the root is present
* Cuspal involovement
* Restoration present

Ages: 4 Years to 7 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Healthy children between ages of four and seven years will be included in this study
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2021-11-01 (Actual); Primary Completion 2022-04-01 (Actual); Study Completion 2022-05-01 (Actual)

PRIMARY OUTCOMES:
healing | 3 months post-operatively
  The assessment of all restorations will be carried out at 24-hours operatively under normal clinical conditions with a dental operating light, a mouth mirror and a dental explorer.
healing | 3 months post-operatively
  The assessment of all restorations will be carried out at 3 months operatively under normal clinical conditions with a dental operating light, a mouth mirror and a dental explorer.
healing | 6 months post-operatively
  The assessment of all restorations will be carried out at 6 months operatively under normal clinical conditions with a dental operating light, a mouth mirror and a dental explorer.

SECONDARY OUTCOMES:
impact of colour | 24-hours, 3, 6 months post-operatively
  assessed once through a questionnaire given to the child at the beginning of the first dental visit in which each child will be asked to choose from pictures that indicate their preference regarding the use of colored and non-colored restorative materials and how their choice will affect their attitude whether they will be happy, sad or neutral.
impact of colour | 3 months post-operatively
  assessed once through a questionnaire given to the child at the beginning of the first dental visit in which each child will be asked to choose from pictures that indicate their preference regarding the use of colored and non-colored restorative materials and how their choice will affect their attitude whether they will be happy, sad or neutral.
impact of colour | 6 months post-operatively
  assessed once through a questionnaire given to the child at the beginning of the first dental visit in which each child will be asked to choose from pictures that indicate their preference regarding the use of colored and non-colored restorative materials and how their choice will affect their attitude whether they will be happy, sad or neutral.

CONTACTS AND LOCATIONS:
Locations (1):
- the British University in Egypt, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No